CLINICAL TRIAL: NCT00412126
Title: Does Reduction of Hyperglycemia With Insulin Impact Restenosis and Improve Clinical Outcomes Following PCI?
Brief Title: Clinical and Angiographic Outcomes With Hyperglycemic Control Post PCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hamilton Health Sciences Corporation (Other)
Collaborators: Heart and Stroke Foundation of Canada (Other)
Organization: McMaster University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 01-223
Record Dates: First submitted 2006-12-13; First posted 2006-12-15 (Estimated); Last update posted 2006-12-15 (Estimated); Status verified 2006-12

CONDITIONS: Diabetes Mellitus; Coronary Restenosis
Keywords: Diabetes Mellitus; Coronary Restenosis; Insulin; Angioplasty
MeSH Terms: conditions — Diabetes Mellitus; Coronary Restenosis; Insulin Resistance | interventions — Insulin

INTERVENTIONS:
Drug: Insulin

SUMMARY:
Coronary artery disease is a process that results in "hardening of the arteries". When the arteries that supply blood and oxygen to your heart muscle become clogged or narrowed, a heart attack may result, or you may feel chest discomfort (angina) - sometimes even while resting. One approach to treating this condition is a balloon procedure known as coronary angioplasty.

The major limitation of coronary angioplasty is renarrowing of the artery (restenosis) in the first six months following the procedure requiring either repeat angioplasty or referral for bypass surgery. Patients with diabetes have always been identified as having higher rates of restenosis and poor outcomes following angioplasty, despite some important scientific advances. We think that the level of blood sugar control at the time of angioplasty and in the following months may be related to the extent of restenosis.

We expect that a reduction in blood sugar with insulin may, in turn, reduce the restenosis process and improve your long-term outcome.

DETAILED DESCRIPTION:
Studies consistently show that diabetes (DM) is an independent predictor of angiographic restenosis as well as clinical outcomes after PCI. A common criticism of the early PCI trials is that stents were not routinely used. However, even when stents are used, the presence of DM is associated with a higher restenosis rate and lower event rate survival. In a series of 3,554 consecutive patients (715 DM patients) undergoing stenting procedures at a single centre the incidence of restenosis and total vessel occlusion by angiographic assessment was significantly higher in diabetes. Increased restenosis rates were consistently demonstrated across a broad range of lesion types.

The pathophysiology of restenosis is viewed as a complex temporal sequence of interactions involving several cellular and mechanical factors including elastic recoil, thrombosis, intimal hyperplasia, extra cellular matrix elaboration, apoptosis, oxidative stress and unfavorable arterial remodeling ("arterial shrinkage"). The exposure of subendothelial elements initiates platelet adhesion and activation. Activated platelets at the site of injury secrete growth factors that release smooth muscle cells from growth inhibition and induce their proliferation and subsequent migration from the media to the intima. Smooth muscle cell proliferation continues beyond the phase of platelet deposition. Extracellular matrix is produced and secreted by smooth muscle cells that have migrated into the injured intimal zone. This hypocellular matrix material forms the bulk of the intimal tissue. Although mechanical factors such as early vessel elastic recoil may play a major role following balloon angioplasty, this mechanism should not significantly affect the stented segments as the stent provides a rigid endovascular scaffold. Similarly, late arterial remodelling which has been postulated to be a significant factor for the development of restenosis after PCI should not have a major effect in the context of stents. Therefore, the major mechanism contributing to in-stent restenosis is aggressive intimal hyperplasia.

Recent studies demonstrate that DM is characterized by diffuse intimal hyperplasia within the stented segment. DM is an independent predictor of the volume of intimal hyperplasia within the stent. The pattern of stent restenosis in patients with DM tends to be more diffuse and proliferative and therefore more likely to lead to total vessel occlusion. This is significant because diffuse restenosis is difficult to manage with repeat percutaneous procedures.

Hyperglycemia has been postulated to promote the restenotic process in diabetes by the following mechanisms: i. endothelial cell dysfunction; ii. increased platelet aggregation and thrombus formation; iii. dysregulation of growth factor expression; iv. abnormal extracellular matrix deposition; v. advanced isolation and products.

Approaches to preventing stent restenosis have had limited effect. Pharmacologic trials have universally failed to show a reduction in restenosis rates in human subjects. Recent reports suggested radiation therapy (brachytherapy) especially applied locally either via catheters or through radioactive stents has a potential to reduce the proliferative response. Although this approach holds great promise there are unresolved logistic issues, safety issues, and cost issues limiting wide-spread application.

Preliminary studies of drug-eluting stents show initial promise in reducing restenosis rates. However, stent coatings can counteract the restenotic process only at points where the stent strut opposes the arterial wall and have little effect on neointimal tissue that can protrude between the struts and into the lumen. Furthermore, both brachytherapy and stent coatings only apply to the stented segments and the vessel whereas the arterial responses to balloon injury may also depend on flow characteristics (i.e. rheology) of the vessel. Therefore, alternative strategies that impact both local processes of the dilatation site and systematic processes on vessel remodelling and rheology are needed.

Clinical trial data suggests that glycemic control may prevent restenosis. A recent study of patients with type 2 diabetes undergoing PCI with stent demonstrated a significant reduction in both neointimal area and neointimal index among participants randomized to the glucose-lowering agent troglitazone. Observational data from two registry studies indicate that diabetic patients with well-controlled hemoglobin A1c had lower rates of restenosis.

Several lines of evidence suggest that insulin is safe and effective in controlling diabetes as well as reducing cardiovascular events. The recently published DIGAMI Study in which patients with myocardial infarction were randomized to an insulin infusion followed by at least three months of intensified insulin therapy showed a 31% reduction mortality in patients receiving intensified therapy. Subcutaneous insulin has been safely used to treat diabetes for almost 80 years. Patients can easily learn to both inject and titrate insulin response to home capillary glucose measurements. Greater than 85% of patients with type II diabetes who were started on insulin can achieve safe and effective metabolic control with one injection per day.

Intravascular ultrasound is the most direct and sensitive technology available for measurement of intravascular hyperplasia volume within the stent. It is the technology that is most likely to uncover a benefit of insulin in reducing restenosis if one exists. This methodology will allow the research question to be answered with the smallest possible sample size. Recent studies demonstrate that detailed cross-sectional analysis of intracoronary stents during motorized IVUS catheter pullback is feasible with excellent reproducibility, safety and can be stored for off-line analysis. Establishing a mechanistic link between glycemic control and restenosis will support the design of larger clinical studies evaluating clinical outcomes.

Primary Study Question

* Does intensive control of glucose levels with insulin in patients with DM reduce volume of intimal hyperplasia within the stented segment as evaluated by intravascular ultrasound (IVUS) at 6 months? Secondary Study Question
* Does intensive glycemic control with insulin reduce restenosis as evaluated by quantitative coronary angiography (QCA) at 6 months
* Does intensive glycemic control with insulin prevent clinical events such as hospital admission for unstable angina and for congestive heart failure, myocardial infarction, stroke, revascularization (PCI, CABG) and death at 12 months.

Primary Hypothesis:

·Intensive glycemic control with insulin in diabetic (DM) patients reduces intimal hyperplasia within the stented segment after percutaneous coronary revascularization

Secondary Hypothesis:

* The reduction in intimal hyperplasia is related to the degree of glycemic control (i.e. HbA1c values); and
* Event-free survival is improved in patients treated with insulin

ELIGIBILITY:
Inclusion Criteria:

1. Patients booked for catheter-based revascularization with balloon angioplasty and coronary stent placement
2. Type II diabetes mellitus
3. On 0-2 oral glucose lowering agents and able to double the dose of (or add) at least one glucose lowering agent. If HbA1c is 0.100-0.104, then must be on only 0-1 oral antidiabetic agents (the dose of one agent must be ≤ ½ max dose) and able to take metformin (i.e. no previous intolerance; and serum creatinine < 130 mol/L)

Exclusion Criteria:

1. Planned staged procedure for multivessel PCI taking place over > 30 days
2. Estimated LVEF < 35%, if known
3. NYHA class 3 or 4 symptoms of CHF
4. HbA1c < 0.061 or > 0..104.
5. Current or anticipated need for insulin or TZD within the next 6 months
6. On > 50% of the maximum doses of an insulin secretagogue and unable to take metformin because of previous intolerance, or because of a serum creatinine  130 mol/L
7. Refusal to take insulin
8. Refusal to do home glucose monitoring
9. History of hypoglycemia requiring 3rd party assistance in the last 2 years
10. Noncardiac illness expected to limit survival.
11. Renal insufficiency (participants not on metformin  creatinine > 180 mol/L; participants on metformin  creatinine > 130 mol/L)
12. Known hepatic disease (ALT > 2 X ULN, if known)
13. Suspected or known pregnancy
14. Refusal/unable to return for follow-up.
15. Enrolled in a competing randomized trial or clinical study.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240
Dates: Start 2002-07; Study Completion 2005-09

PRIMARY OUTCOMES:
Volume of intimal hyperplasia in the stented segment by IVUS at 6 months following PCI

SECONDARY OUTCOMES:
Late loss in minimal luminal diameter of stented site in coronary vessel evaluated by QCA at 6 months post-PCIb) Rate of clinical events at one year (hospital admission for unstable angina, CHF, MI, stroke, revascularization, and death)

CONTACTS AND LOCATIONS:
Overall Officials: Madhu K Natarajan, MD, FRCPC, Principal Investigator — Hamilton Health Sciences Corporation
Locations (1):
- McMaster University/Hamilton Health Sciences, Hamilton, Ontario, Canada

REFERENCES:
- [Derived] Natarajan MK, Strauss BH, Rokoss M, Buller CE, Mancini GB, Xie C, Sheth TN, Goodhart D, Cohen EA, Seidelin P, Harper W, Gerstein HC. Randomized trial of insulin versus usual care in reducing restenosis after coronary intervention in patients with diabetes. the STent Restenosis And Metabolism (STREAM) study. Cardiovasc Revasc Med. 2012 Mar-Apr;13(2):95-100. doi: 10.1016/j.carrev.2011.12.001. Epub 2012 Jan 30. PMID 22296781